CLINICAL TRIAL: NCT03860948
Title: A Randomized, Open-label, Crossover Pharmacokinetic and Bioequivalence Study of Savolitinib Tablets Produced by Two Different Processes in Healthy Chinese Male Volunteers
Brief Title: A Pharmacokinetic and Bioequivalence Study of Savolitinib Tablets in Healthy Chinese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-504-00CH1
Record Dates: First submitted 2019-02-25; First posted 2019-03-04 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-02

CONDITIONS: Bioequivalence
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Savolitinib Test Preparation (Experimental): The subjects in this arm will receive Test preparation (T). T is dry granulation savolitinib tablets.
  Interventions: Drug: Savolitinib Test Preparation
- Savolitinib Reference Preparation (Experimental): The subjects in this arm will receive Reference preparation(R). R is wet granulation savolitinib tablets.
  Interventions: Drug: Savolitinib Reference Preparation

INTERVENTIONS:
Drug: Savolitinib Test Preparation — Test preparation (T): dry granulation savolitinib tablets.
  Other Names: HMPL-504, volitinib, AZD6094
  Arms: Savolitinib Test Preparation
Drug: Savolitinib Reference Preparation — Reference preparation (R): wet granulation savolitinib tablets.
  Other Names: HMPL-504, volitinib, AZD6094
  Arms: Savolitinib Reference Preparation

SUMMARY:
This is a single-center, randomized, open lebal, single-dose, three-period, crossover clinical study in healthy Chinese male subjects to assess the pharmacokinetics and bioequivalence/bioavailability of two formulation savolitinib tablets.

DETAILED DESCRIPTION:
Thirty six Chinese male subjects who met the inclusion criteria but not met the exclusion criteria, will be hospitalized in Phase I Ward one day before first dosing and randomized into three groups, 12 subjects each, at a ratio of 1:1:1. The subjects in the different group will follow the fixed dosing regimen with 600 mg savolitinib tablets (200 mg/tablet x 3 tablets) after the standard meal on day 1 in cycle 1, 2 and 3 respectively: TRR, RTR or RRT, where "T" indicates dry granulation savolitinib tablet and "R" indicates wet granulation savolitinib tablet. PK blood samples, 2 mL each time, will be collected at the following time points in each dosing cycle: within 0.5 hours before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48 hours after dosing(16 time-points).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must agree to comply with the protocol and Informed consent must be obtained in writing for all subjects;
2. Healthy male subjects aged 18 to 45 years inclusive at the time of screening;
3. Weight ≥ 50 kg, body mass index (BMI) of 19-26 kg/m2;
4. No clinically significant abnormalities or findings in medical history, vital signs, physical examination, 12-lead ECG and laboratory values;
5. Males with the ability to have children must commit to adopting reliable contraceptive measures (e.g. condoms, contraceptive sponges, contraceptive gels, contraceptive films, intrauterine devices, contraceptives for oral or injectable intake, subcutaneous implants or other contraceptives) in collaboration with their partners for the duration of the study and for three months after the final dosage.

Exclusion Criteria:

1. History or symptoms of a clinically significant illness in metabolic/ endocrine, liver, kidney, blood, lung, immune system, cardiovascular, gastrointestinal, genitourinary, neurological, or psychiatric systerm in the 3 months before the study, as determined by the investigator;
2. History of gastrointestinal surgery, kidney surgery and cholecystectomy, which may potentially affect the absorption or excretion of drugs, as determined by the investigator ;
3. History of a severe allergy (for example, certain drug allergy) and acute allergic rhinitis or food allergy within 2 weeks prior to the screening stage;
4. Serum albumin < 35 g/L;
5. Hypertention: systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg
6. Mean corrected QT interval (QTcF) in electrocardiograms (ECG), males > 450 milliseconds, or existing factors that may increase the risk of QTc prolongation, such as chronic hypokalemia that cannot be corrected by potassium supplementation, or congenital or familial long QT syndrome or a family history of unexplained sudden death under 40 years of age in first-degree relatives, or use any combination of drugs known to prolong the QT interval and cause torsades de pointes.
7. Clinical significant abormal findings in Chest X-ray (posteroanterior position) examination;
8. Serum virology positive findings, including HBS Ag, HCV Ab, HIV Ab, or TP Ab;
9. Current smoker of more than 10 cigarettes or equivalent / day during past 3 month prior to commencing the study and unable to completely stop smoking during the study;
10. Have blood or blood products transfusion within 2 months; or blood donation of more than 250 mL within 1 month or 400 mL within 3 months prior to screening; or planning to donate blood or blood components during the study or within 1 month after the end of the study;
11. History of alcohol abuse or drug addiction within one year prior to screening;
12. Participation in any other investigational drug clinical study while last dose was administrated within three months prior to the screening.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
The area under the curve(AUC) of savolitinib | Measured on the Cycle1 Day1 to Day3, Cycle2 Day1 to Day3, Cycle3 Day1 to Day3, each cycle is 10 days.
  The area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration.
Maximum observed plasma concentration (Cmax) of savolitinib | Measured on the Cycle1 Day1 to Day3, Cycle2 Day1 to Day3, Cycle3 Day1 to Day3, each cycle is 10 days.
  Maximum observed concentration, occurring at Tmax.
The time to Cmax (peak time, Tmax) of savolitinib | Measured on the Cycle1 Day1 to Day3, Cycle2 Day1 to Day3, Cycle3 Day1 to Day3, each cycle is 10 days.
  The time at which maximum plasma concentration (Cmax) is observed.
Half-life (t1/2) of savolitinib | Measured on the Cycle1 Day1 to Day3, Cycle2 Day1 to Day3, Cycle3 Day1 to Day3, each cycle is 10 days.
  The time required for the concentration of the drug to reach half of its original value.
Bioequivalence of savolitinib | Measured on the Cycle1 Day1 to Day3, Cycle2 Day1 to Day3, Cycle3 Day1 to Day3, each cycle is 10 days.
  A term in pharmacokinetics used to assess the expected in vivo biological equivalence of two proprietary preparations of a drug.

SECONDARY OUTCOMES:
To observe the safety of healthy volunteers after a single oral dose of savolitinib | From the first dose to within 12 days after the last dose
  Incidence of adverse events evaluated by NCI CTCAE v4.03
Relative bioavailability of savolitinib | Measured on the Cycle1 Day1 to Day3, Cycle2 Day1 to Day3, Cycle3 Day1 to Day3, each cycle is 10 days.
  The area under the curve (AUC) is the definite integral in a plot of drug concentration in blood plasma vs. time.

CONTACTS AND LOCATIONS:
Overall Officials: Jingying Jia, Principal Investigator — Shanghai Xuhui District Central Hospital
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No